CLINICAL TRIAL: NCT01793051
Title: A Phase II Randomized Study of the Efficacy of Minocycline vs. Placebo to Reduce Symptom Burden During Maintenance Therapy for Multiple Myeloma
Brief Title: Intervention for Symptom Burden During Maintenance Therapy for Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012-0413; P01CA124787 (NIH); NCI-2013-00700 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2013-02-13; First posted 2013-02-15 (Estimated); Results first posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Myeloma
Keywords: Myeloma; Multiple Myeloma; MM; Symptom Burden; Symptom reduction; Maintenance therapy with lenalidomide; Minocycline; Dynacin; Minocin; Minocin PAC; Myrac; Solodyn; Placebo; Sugar pill; MD Anderson Symptom Inventory; MDASI; Questionnaires; Surveys
MeSH Terms: conditions — Neoplasms, Plasma Cell; Multiple Myeloma; cyclopia sequence | interventions — Minocycline; Sugars; Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Minocycline (Experimental): Minocycline 200 mg by mouth for the first dose, then 100 mg by mouth every 12 hours for three months beginning at initiation of Lenalidomide maintenance chemotherapy for MM.
  Completion of MD Anderson Symptom Inventory (MDASI) questionnaires at baseline, weekly during Lenalidomide therapy, and at end of treatment visit.
  Interventions: Drug: Minocycline; Behavioral: Questionnaires
- Placebo (Placebo Comparator): Placebo 200 mg by mouth for the first day of Lenalidomide maintenance therapy for MM, then 100 mg doses every 12 hours for three months (three cycles of maintenance chemotherapy).
  Completion of MD Anderson Symptom Inventory (MDASI) questionnaires at baseline, weekly during Lenalidomide therapy, and at end of treatment visit.
  Interventions: Other: Placebo; Behavioral: Questionnaires

INTERVENTIONS:
Drug: Minocycline — 200 mg by mouth for the first dose, then 100 mg by mouth every 12 hours for three months beginning at initiation of Lenalidomide maintenance therapy for MM.
  Other Names: Dynacin; Minocin; Minocin PAC; Myrac; Solodyn
  Arms: Minocycline
Other: Placebo — 200 mg by mouth for the first day of Lenalidomide maintenance therapy for MM, then 100 mg doses every 12 hours for three months (three cycles of maintenance chemotherapy).
  Other Names: Sugar pill
  Arms: Placebo
Behavioral: Questionnaires — Completion of MD Anderson Symptom Inventory (MDASI) questionnaires at baseline, weekly during Lenalidomide therapy, and at end of treatment visit.
  Other Names: Surveys; MD Anderson Symptom Inventory; MDASI

SUMMARY:
The goal of this clinical research study is to learn if minocycline can help reduce the symptoms reported by patients with MM who receive therapy with lenalidomide.

Minocycline is an antibiotic and has been shown to interrupt pro-inflammatory cytokine production, which may help to reduce multiple symptoms.

DETAILED DESCRIPTION:
Study Groups:

If participant agrees to take part in this study, they will be randomly assigned (as in the flip of a coin) to 1 of 2 groups.

Group 1 will take a placebo during maintenance therapy.

Group 2 will take minocycline during maintenance therapy.

A placebo is not a drug. It looks like the study drug but it is not designed to treat any disease or illness. It is designed to be compared with a study drug to learn if the study drug has any real effect.

Neither participant nor the study staff will know if participant is receiving the study drug or the placebo. However, if needed for participant's safety, the study staff will be able to find out what they are receiving.

Study Drug Administration:

Participant will take the study drug/placebo by mouth, two times a day for about 3 months, starting the first day (or within 2 days) that they begin their lenalidomide therapy.

Participant should take the study drug/placebo with a full glass (8 ounces) of water. Participant may take it with or without food, but if the study drug/placebo causes an upset stomach, participant should take it with food.

Study Visits:

Participant must bring the study drug/placebo container, along with any remaining drug, with them to their clinic visit at each new cycle of lenalidomide therapy, or at the clinic visit when the study is over if no clinic visits are scheduled until then.

Before participant starts lenalidomide therapy:

* Participant will fill out 4 questionnaires about pain and other symptoms. It should take about 20-25 minutes to complete all of the questionnaires.
* A study staff member will ask participant questions about their demographic information, such as their marital status, job status, education, and race.
* Blood (about 2 tablespoons) will be drawn for biomarker testing. This will be during an already scheduled blood draw and participant would not need to have an extra needle stick. Biomarkers are found in the blood/tissue and may be related to participant's reaction to the study drug. Researchers want to study how changes in the biomarkers may be related to the symptoms reported by participants in this study.

During lenalidomide therapy:

°Participant will complete a symptom questionnaire in the clinic or by telephone 1 time each week about any symptoms they may be having and how they may be affecting participant's daily activities. The symptom questionnaire should take about 3-5 minutes to complete each time.

During participant's clinic visit at each new cycle of lenalidomide therapy:

* Participant will fill out 3 questionnaires about their pain and other symptoms. It should take about 15-20 minutes to complete all of the questionnaires each time. If no clinic visit is scheduled until the study is over, these questionnaires will be collected over the phone by the study coordinator.
* Blood (about 2 tablespoons) will be drawn for biomarker testing. This will be during an already scheduled blood draw and participant would not need to have an extra needle stick.

End-of-Treatment Visit:

Participant will have an end-of-treatment visit at the end of month 3. At this visit, participant will complete 4 questionnaires about pain and other symptoms. It should take about 20-25 minutes to complete all of the questionnaires. Blood (about 2 tablespoons) will be drawn for biomarker testing. This will be during an already scheduled blood draw and participant would not need to have an extra needle stick.

Length of Study:

Participant may continue taking the study drug/placebo for up to 3 months. Participant will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, if they are unable to follow study directions, or the study doctor thinks it is in their best interest.

This is an investigational study. Minocycline is FDA approved and commercially available for the treatment of bacterial infection. The use of minocycline to reduce chemotherapy related side effects in patients with MM is currently being used for research purposes only.

Up to 88 participants will take part in this study. All will be enrolled at MD Anderson Cancer Center.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with pathologically diagnosed who have received induction chemotherapy, with or without AuSCT, and who have qualified to receive lenalidomide-based maintenance therapy for their MM.
2. Patients > or = 18 years old.
3. Patients able to render informed consent and to follow protocol requirements.
4. Patients who speak English (due to patient-reported outcome language options, we are only accruing English-speaking patients to the protocol).
5. Patients with normal renal function according to MD Anderson testing standards and no prior renal disease [screening cut off for serum creatinine < 1.5 times the upper limit of normal].
6. Patients with normal hepatic function according to MD Anderson testing standards and no prior liver disease [screening results for total bilirubin must be < 1.5 times the upper limit of normal; screening results for alkaline phosphatase (ALP) and alanine aminotransferase (ALT) must be < 2 times the upper limit of normal; if available, screening results for aspartate aminotransferase (AST) must be < 2 times the upper limit of normal].

Exclusion Criteria:

1. Patients who are taking minocycline for other conditions, as determined by the treating physician
2. Patients with hypersensitivity to tetracyclines
3. Women who are pregnant or nursing; pregnancy will be confirmed by urine test
4. Patients who are enrolled in other clinical trials that have symptom management as primary outcome
5. Patients who are not able to use telephone-based interactive voice response software due to physical limitations (e.g., impaired hearing)
6. Patients taking any tetracycline in the last 15 days
7. Patients on Vitamin K antagonist warfarin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2013-03-22 (Actual); Primary Completion 2020-09-18 (Actual); Study Completion 2020-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Orlowski, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All recruitment done at the University of Texas MD Anderson Cancer
Pre-assignment Details: 88 participants enrolled and randomized to either the intervention group or the control group. 1 patient withdrew before the study began.
Groups:
- Minocycline: Minocycline 100 mg (capsule) two times a day to begin with start of maintenance therapy (3 months +/- 2 days)
- Placebo: Placebo 100 mg (capsule) two times a day to begin with start of maintenance therapy (3 months +/- 2 days)
Period: Overall Study
Arm/Group | Minocycline | Placebo
Started | 43 | 44
Completed | 33 | 36
Not Completed | 10 | 8
Not completed — Withdrawal by Subject | 6 | 4
Not completed — Adverse Event | 0 | 2
Not completed — Too ill to continue | 1 | 0
Not completed — Switched chemo | 1 | 1
Not completed — Lack of compliance | 1 | 0
Not completed — Requested to be removed from the study | 1 | 1

BASELINE CHARACTERISTICS:
Population: Evaluable participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Minocycline | Placebo | Total
Number analyzed (Participants) | 33 | 36 | 69
Age, Continuous [Mean (Full Range); unit: years] | 62 [44 to 72] | 60 [46 to 81] | 61 [44 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 7 | 18
  Male | 22 | 29 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 26 | 27 | 53
  Unknown or Not Reported | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  United States | 33 | 36 | 69

OUTCOME MEASURES:

1. Primary Outcome: Symptom Reduction
Description: Minocycline tested for its ability to reduce the value of a patient's 3 month (± two days) area under the curve (AUC) for the mean of 5 symptoms: fatigue, pain, muscle weakness, numbness, and bone aches. The AUC is calculated using a trapezoidal approximation, derived by multiplying half of the base with the sum of the two heights. The two heights correspond to the two mean symptom scores computed at each of these assessments. The AUC is measured in units of mean MDASI score in days. The area for the subsequent trapezoid can be calculated in the same way. Given a baseline, weekly assessment schedule over a three month period and end of trial assessment, there will be a total of 14 trapezoids. The AUC is the sum of the area of the 14 trapezoids. Each of the trapezoid has a maximum value of 70 (0.5*7 days*(10+10)). Hence, the AUC will have a minimum score of 0 and a maximum score of 980. Higher AUC values indicate worse outcomes.
Time Frame: Baseline to 3 months (three cycles with assessments made at beginning of each)
Measure: Mean (Standard Deviation); unit: units on a scale*month
Arm/Group | Minocycline | Placebo
Number analyzed (Participants) | 33 | 36
units on a scale*month | 26.02 (17.72) | 26.65 (21.19)

ADVERSE EVENTS:
Time Frame: From the start of the study medication, up to 30 days after last dose administered, up to a total of 4 months
Arm/Group | Minocycline | Placebo
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/36
Other Adverse Events (participants affected / at risk) | 3/33 | 4/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Minocycline (N=33) | Placebo (N=36)
Anxiety (Nervous system disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Blurred Vision (Eye disorders) | 1 | 3
Constipation (Gastrointestinal disorders) | 2 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cytopenia (Blood and lymphatic system disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 2
Dizziness (Nervous system disorders) | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-07): https://cdn.clinicaltrials.gov/large-docs/51/NCT01793051/Prot_SAP_000.pdf